CLINICAL TRIAL: NCT03992391
Title: Developing and Implementing an Adolescent Suicide Prevention Program in a Community Mental Health Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Beth Kennard, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 112016-061
Record Dates: First submitted 2019-01-02; First posted 2019-06-20 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Phase 1: Treatment Development Phase 2: Pilot Group Phase 3: Open Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qualitative Interviews (No Intervention): Qualitative Interviews with adolescents, their parents and clinicians.
- Open Pilot (Experimental): Open-label pilot group of adolescents (n=10) in a suicide prevention intensive outpatient program
  Interventions: Behavioral: Suicide Prevention Intensive Outpatient Program
- Open-label trial (Experimental): Open-label trial of adolescents (n=40) in a suicide prevention intensive outpatient program
  Interventions: Behavioral: Suicide Prevention Intensive Outpatient Program

INTERVENTIONS:
Behavioral: Suicide Prevention Intensive Outpatient Program — participation in a suicide prevention intensive outpatient program
  Arms: Open Pilot; Open-label trial

SUMMARY:
This is a three phase study to develop and implement an adolescent suicide prevention program in a community mental health setting. In Phase 1, needs assessments using qualitative interviews will be conducted at in a community mental health clinic with suicidal teens and their parents, and with community experts including therapy staff who serve patients at a community mental health clinic. In Phase 2, the investigators will develop a new treatment manual that is guided by information obtained in the previously completed needs assessment. The investigators will pilot the program with one group of adolescents (N=10), and make iterative revisions based on feedback. Training sessions will be implemented. In Phase 3, the investigators will conduct an open trial of a group for 40 adolescents at the community mental health clinic to assess feasibility of recruitment, implementation, satisfaction, and outcome. Program outcomes will be utilization, patient and family satisfaction ratings, and improvement in depression and suicide risk measures at discharge from the program and at one month and six months follow-up. In addition, rate of suicidal events (suicide attempt, hospitalization) at one month and six months post-discharge will be compared to historical controls.

DETAILED DESCRIPTION:
In Phase 1, the investigators will develop interviews and data collection guides. The investigators will interview 10 current patients and parents at a community mental health clinic (for a total of 20 individuals). The investigators will elicit respondent perspectives relating to: (a) utilization of care (b) treatment targets (c); parent/family participation and (d) session format. Also, as part of Phase 1, the investigators will conduct interviews with the 8 treatment providers at a community mental health clinic. In addition to exploring the content of treatment modules of the intensive outpatient program (IOP) program, the investigators will share responses from patients and parents, and will solicit provider feedback regarding those responses. Building on patient-reported needs, the investigators will solicit provider expectations, requisite elements and other concerns regarding implementation of an intensive treatment program in community mental health clinic settings. Coders will independently read the transcripts and code for common elements. Developing a codebook to document procedures, the investigators will compare and contrast codes and respective quotations across respondents. Coding discrepancies will be discussed and conflicts between raters resolved using a third investigator. The investigators will present the preliminary manual content to clinician respondents to explore feasibility of the proposed intervention. Data will be coded and analyzed using standard qualitative approaches and will guide the manual development and intervention components to be used in Phases 2 and 3.

In Phase 2, the investigators will incorporate responses into a draft of treatment manual, and train a group of community mental health clinic staff to deliver treatment. The investigators will test this adapted manual with an open trial to test feasibility and piloting of the intervention and outcome measures. Patients and parents will complete the Quick Inventory of Depressive Symptomatology - Adolescents (QIDS-A). Client Satisfaction Questionnaire (CSQ) will be obtained at discharge. Participants will complete the Interpersonal Needs Questionnaire (INQ), Concise Health Risk Tracking (CHRT) , and the Acquired Capability for Suicide Scale (ACSS) at both intake and discharge, Clinicians will complete the Clinician Checklist and the Columbia Suicide Severity Rating Scale (C-SSRS) at baseline and discharge. The investigators will conduct exit interviews completed with both the parent and patient, to assess the acceptability of treatment. The investigators will obtain feedback about perceived effectiveness of the treatment, the appropriateness of treatment targets, identification of other targets or approaches that would have been more helpful, and barriers to participation. The investigators will obtain similar feedback from the treating clinicians. Based on patient, family, and clinician feedback, a satisfaction questionnaire (patient and parent), and outcome data from the open trial, the manual, treatment program structure can be modified in Phase 3 to improve feasibility and acceptability. The investigators will collect follow-up information at 1 month and 6 months following the patient's final session.

In Phase 3, participants will be 40 adolescents who present to the community mental health clinic with a recent suicide attempt or significant suicidal ideation with a plan or intent. Participants must be English-speaking, although parents must be able to speak Spanish. Participants can have unipolar or bipolar disorder, conduct or oppositional disorder, eating disorder, or alcohol or substance use or abuse, all of which are common comorbidities in the suicidal adolescent sample. Excluded are those with current psychosis, mania, alcohol or substance dependence, autism spectrum disorders, <80% of ideal body weight, or low intelligence quotient (IQ) based on clinical judgement (if concerns about intellectual capabilities are evident at assessment), as these conditions may require more intensive interventions or limit comprehension of the intervention components. The program will include 1-2 hours of group therapy once weekly, and utilize Cognitive Behavioral Therapy and Dialectical Behavior Therapy components focusing on skills to reduce risk factors associated with suicidal behaviors. The selection and emphasis on specific skills will be based on input during the early phases of the project. Length of treatment is expected to be 6-8 weeks, depending on individual patient need. Adolescents also will receive individual and/or family therapy, and will be referred to a psychiatrist for medication management as needed. In addition, parents will attend a 1-hour biweekly skills-based parent group.

Outcome Measures. Patients and parents will complete the Quick Inventory of Depressive Symptomatology - Adolescents (QIDS-A). Client Satisfaction Questionnaire (CSQ) will be obtained at discharge. Participants will complete the Interpersonal Needs Questionnaire (INQ), Concise Health Risk Tracking (CHRT), and the Acquired Capability for Suicide Scale (ACSS) at both intake and discharge, Clinicians will complete the Clinician Checklist and the Columbia Suicide Severity Rating Scale (C-SSRS) at baseline and discharge. The investigators will collect follow-up information at 1 month and 6 months following each patient's final session.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying Latino/Latina adolescents (aged 12-17 years) currently in outpatient treatment at Metrocare and who struggle with depression and/or suicidal ideations
* Adolescents must speak English fluently as the self-report forms do not have normative data for non-English speaking subjects, and the confidential nature of therapy prevents us from being able to use a translator for visits. Parents of participants may speak Spanish or English.

Exclusion Criteria:

* current psychosis
* mania
* alcohol or substance dependence
* autism spectrum disorders
* <80% of ideal body weight
* IQ<70 (based on clinical judgement)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Adolescents (QIDS-A) | through program completion, an average of 6 weeks
  measure of depression symptom severity, total range = 0-27, lower values are considered to be better (less depressed) than higher values (which indicate more depressed). Lower scores indicate a better outcome than higher scores. No subscales.
Concise Health Risk Tracking (CHRT) | through program completion, an average of 6 weeks
  measure of suicide propensity and risk
Client Satisfaction Questionnaire (CSQ) | at program completion, on average 6 weeks after program completion
  measure of client satisfaction
Follow-up Interview | one-month after program completion
  to assess subsequent suicidal behaviors, service utilization, and ongoing psychiatric and psychosocial treatment adherence

CONTACTS AND LOCATIONS:
Overall Officials: Beth D. Kennard, PsyD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Metrocare Services, Dallas, Texas, United States